CLINICAL TRIAL: NCT05568368
Title: Time-to-Detection in Culture of Mycobacterium Tuberculosis : Performance for Assessing Index Cases Infectivity
Brief Title: Time-to-Detection in Culture of Mycobacterium Tuberculosis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Infectio01
Record Dates: First submitted 2022-10-04; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Tuberculoses
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Index cases
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
determination if time-to-detection in cultures of M. tuberculosis samples is more discriminating than acid-fast staining in transmission

ELIGIBILITY:
Inclusion Criteria:

* have at least 1 contact case explored for tuberculosis
* latent tuberculosis infection

Exclusion Criteria:

-

Ages: 2 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all cases of pulmonary tuberculosis who had a sample analysed by the laboratory of bacteriology of Nice University Hospital, and that was positive in culture before treatment and of which contact cases were explored by the CLAT
Sampling Method: Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
tuberculosis transmission | 2 months
  duration of Tuberculosis transmission between an infected person and a contact case
contact case tracking | 2 months
  screening time for contact cases

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No